CLINICAL TRIAL: NCT06602024
Title: A Phase 3, Randomized, Observer-blind, Active-controlled, Case-driven Study to Investigate the Safety, Efficacy, and Immunogenicity of mRNA-1010 Candidate Seasonal Influenza Vaccine Compared With a Licensed Inactivated Seasonal Influenza Vaccine in Adults ≥50 Years of Age
Brief Title: A Study of mRNA-1010 Compared With a Licensed Influenza Vaccine in Adults ≥50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1010-P304; 2024-516240-26-00 (Other: EU CT)
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Seasonal Influenza
Keywords: Seasonal Influenza; Flu; mRNA-1010; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine; fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1010 (Experimental): Participants will receive a single injection of mRNA-1010 on Day 1.
  Interventions: Biological: mRNA-1010
- Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra (Active Comparator): Participants will receive a single injection of active comparator trivalent influenza vaccine (TIV) or quadrivalent influenza vaccine (QIV) (Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra) on Day 1.
  Interventions: Biological: Fluarix®; Biological: Influsplit® Tetra; Biological: Fluarix Tetra; Biological: Alpharix® Tetra

INTERVENTIONS:
Biological: mRNA-1010 — Intramuscular (IM) injection
  Arms: mRNA-1010
Biological: Fluarix® — IM injection
  Arms: Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra
Biological: Influsplit® Tetra — IM injection
  Arms: Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra
Biological: Fluarix Tetra — IM injection
  Arms: Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra
Biological: Alpharix® Tetra — IM injection
  Arms: Fluarix®, Fluarix Tetra, Influsplit® Tetra, Alpharix® Tetra

SUMMARY:
The primary objectives of this study are to evaluate the safety and reactogenicity of mRNA-1010, and to evaluate relative vaccine efficacy (rVE) of mRNA-1010 versus an active comparator against reverse transcription polymerase chain reaction (RT-PCR)-confirmed protocol-defined influenza-like illness (ILI) caused by any influenza A or B strains.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Participants who are assigned female at birth or can become pregnant are eligible to participate if:

  * The participant is a person of nonchildbearing potential (PONCBP) or
  * The participant is a person of childbearing potential (POCBP) who:
* Is not breast/chest feeding.
* Is using an acceptable contraceptive method at least 28 days prior to Day 1 (Baseline) to at least 90 days after Day 1 (Baseline).
* Has a negative highly sensitive pregnancy test (urine or serum as required by local regulation or institutional review board [IRB]/independent ethics committee [IEC]) at the Screening Visit and before study intervention (if the Day 1 [Baseline] Visit is not on the same day as the Screening Visit).

Exclusion Criteria:

* Acutely ill or febrile (temperature ≥38.0 degrees Celsius (℃) [100.4° Fahrenheit [F]]) within 72 hours prior to Day 1 (Baseline).
* Close contact with someone with laboratory-confirmed influenza infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu®/oseltamivir) within 5 days prior to Day 1 (Baseline).
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of congenital or acquired immunodeficiency, immunosuppressive condition, asplenia, or recurrent severe infections disease.
* Tested positive for influenza by local health authority-approved testing methods within 180 days prior to Day 1 (Baseline).
* History of anaphylaxis or severe hypersensitivity reaction requiring medical intervention after receipt of any of the following: mRNA vaccine or therapeutic; components of an mRNA vaccine or therapeutic; influenza vaccine; or components of an influenza vaccine, including egg protein.
* Malignancy within 2 years prior to Day 1 (Baseline) (adequately treated basal cell carcinoma and squamous cell carcinoma are allowed).
* Received corticosteroids at ≥10 milligram (mg)/day of prednisone or equivalent for >14 days in total within 90 days prior to Day 1 (Baseline) or is anticipating the need for corticosteroids at any time during the study.
* Received systemic immunosuppressive treatment, including long-acting biological therapies that affect immune responses (for example, infliximab), within 180 days prior to Day 1 (Baseline) or plans to do so during the study.
* Treated with antiviral therapies for influenza (for example, Tamiflu) within 180 days prior to Day 1 (Baseline).
* Received any vaccine authorized or approved by local health agency within 28 days prior to Day 1 (Baseline) or plans to do so within 14 days after Day 1 (Baseline).
* Received a licensed seasonal influenza vaccine within 180 days prior to Day 1 (Baseline) or plans to do so (outside of this study) at any time during the study.
* Received an investigational seasonal influenza vaccine within 1 year prior to Day 1 (Baseline). Note: participants from mRNA-1010-P304 Season 1 are NOT eligible to re enroll into Season 2.
* Participated in a clinical study with investigational treatment within 90 days prior to Day 1 (Baseline) based on the medical history interview or plans to do so while participating in this study.
* Is working or has worked as study personnel or is an immediate family member or house member of study personnel, study staff, or Sponsor personnel.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40817 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Day 1 to Day 7
Number of Participants with Unsolicited Adverse Events (AEs) | Day 1 to Day 28
Number of Participants with Medically Attended AEs (MAAEs), AEs Leading to Discontinuation, Serious Adverse Events (SAEs), or Adverse Events of Special Interest (AESI) | Day 1 to Day 181
Time to First Episode of RT-PCR Confirmed Protocol Defined ILI | Day 14 up to End of Season (up to approximately Day 181)
  ILI caused by any influenza A or B strains.

SECONDARY OUTCOMES:
Number of Participants with First Episode of RT-PCR Confirmed Modified US Centers for Disease Control and Prevention (CDC)-Defined ILI | Day 14 up to End of Season (up to approximately Day 181)
  ILI caused by any influenza A or B strains.
Number of Participants with First Episode of RT-PCR Confirmed Protocol-Defined ILI or Modified CDC-Defined ILI | Day 14 up to End of Season (up to approximately Day 181)
  ILI caused by influenza A or B strains with antigenic match to the vaccine strains.
Geometric Mean Titer (GMT) of Hemagglutination Inhibition (HAI) | Day 29
  Humoral immunogenicity.
Number of Participants Reaching Seroconversion as Measured by HAI | Day 29
Number of Participants with an HAI Titer ≥1:40 | Day 29
Geometric Mean Fold Rise (GMFR) of HAI Titers | Day 1, Day 29
HAI Titers | Day 29
  As measured by the HAI Assay.
Number of Participants with First Episode of RT-PCR-Confirmed Protocol-Defined ILI | Day 14 up to End of Season (up to approximately Day 181)
  Correlates of Risk (CoR) and Correlates of Protection (CoP).

CONTACTS AND LOCATIONS:
Locations (301):
- United States (188):
  - Pinnacle Research Group, Llc, Anniston, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - Flourish Research, Birmingham, Alabama
  - EmVenio Research Brimingham, AL, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Optimal Research, Huntsville, Alabama
  - Velocity Clinical Research, Mobile, Alabama
  - Lenzmeier Family Medicine, Glendale, Arizona
  - DM Clinical Research, Phoenix, Arizona
  - Helios Clinical Research, Phoenix, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Woodland Research, Rogers, Arkansas
  - Benchmark Research - Colton, Colton, California
  - Flourish Research, Covina, California
  - Velocity Clinical Research - Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Long Beach Research Institute LLC, Long Beach, California
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - M3 Wake Research/PRI, LLC, Newport Beach, California
  - Carbon Health North Hollywood, North Hollywood, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Paradigm Research, Redding, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - Velocity Clinical Research - Banning, San Bernardino, California
  - Artemis Institute for Clinical Research - Research Site, San Diego, California
  - WHCR- M3 Wake Research, San Diego, California
  - Wr-McCr, Llc, San Diego, California
  - Velocity Clinical Research, Santa Ana, California
  - Diablo Clinical Research, Walnut Creek, California
  - Tekton Research - Fort Collins, Fort Collins, Colorado
  - Tekton Research, Inc - Longmont Center, Longmont, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - JEM Research Institue, Atlantis, Florida
  - Nature Coast Clinical Research, LLC - Crystal River, Crystal River, Florida
  - Homestead Associates in Research,Inc, Hialeah, Florida
  - CenExel RCA, Hollywood, Florida
  - Nature Coast Clinical Research, LLC - Inverness, Inverness, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness INC, Jupiter, Florida
  - M3 Wake Research/MSRA,LLC, Lake City, Florida
  - Accel Clinical Research, Lake Mary, Florida
  - Clinical Site Partners - Leesburg, Leesburg, Florida
  - ARS - Meridien Research, Maitland, Florida
  - K2 medical research, Maitland, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Headlands Research, Orlando, Florida
  - Suncoast Research Associates, Pembroke Pines, Florida
  - Health Awareness INC, Port Saint Lucie, Florida
  - IMA Clinical Research Warren, St. Petersburg, Florida
  - Forward Clinical Trials - Dermatology, Tampa, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - JAVARA, Albany, Georgia
  - IACT Health, Columbus, Georgia
  - CenExel iResearch , LLC, Decatur, Georgia
  - CenExel iResearch Savannah, Savannah, Georgia
  - Velocity Clinical Research-Savannah, Savannah, Georgia
  - Javara - Privia Medical Group Georgia, LLC, Savannah, Georgia
  - Clinical Research Atlanta/Headlands, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - EmVenio Research, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - DM Clinical Research- River Forest, Melrose Park, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research-Sioux City, Sioux City, Iowa
  - Alliance for Multispecialty Research, Augusta, Kansas
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - DelRicht Research - Overland Park, Overland Park, Kansas
  - AMR, Wichita, Kansas
  - Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - IMA Clinical Research Monroe, Monroe, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Velocity Clinical Research, New Orleans, Louisiana
  - DelRicht Research @ Neighborhood Health, Prairieville, Louisiana
  - Privia Medical Group, Annapolis, Maryland
  - Cenexel CBH (CBH Health), Gaithersburg, Maryland
  - Matthew Mintz Clinic, Rockville, Maryland
  - Velocity Clinical Research - Covington, Rockville, Maryland
  - DM Clinical Research - Brookline, Brookline, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research, Southfield, Michigan
  - DELRICHT RESEARCH at GULFPORT MEMORIAL, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinvest, Springfield, Missouri
  - Delricht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Delricht, Town and Country, Missouri
  - Boeson Research MSO, Missoula, Montana
  - Elias Research Associates, Missoula, Montana
  - Velocity Clinical Research-Grand Island, Grand Island, Nebraska
  - Platinum Research Network, LLC, Lincoln, Nebraska
  - Velocity Clinical Research-Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research-Omaha, Omaha, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - M3 Wake Research/CRCN, LLC, Las Vegas, Nevada
  - Office of Michael B. Jacobs, MD, Las Vegas, Nevada
  - DM Clinical Research - New Jersey, Jersey City, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - DM Clinical Research-Albuquerque, Albuquerque, New Mexico
  - AXCES Research Group - Sante Fe, Albuquerque, New Mexico
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - DM Clinical, Brooklyn, New York
  - RCR Buffalo, Buffalo, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - IMA Clinical Research, Hartsdale, New York
  - IMA Research, New York, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Velocity Clinical Research-Vestal, Vestal, New York
  - Asheville Clinical Research, Asheville, North Carolina
  - DelRicht Research, LLC, Charlotte, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Eximia Clinical Research, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare US Inc., Salisbury, North Carolina
  - Accellacare Research Wilmington, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Javara - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Velocity Clinical Research-Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Centricity Research Columbus, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Tekton Research, Inc - Edmond, Edmond, Oklahoma
  - Delricht Tate, Tulsa, Oklahoma
  - Tekton Research, Inc - Yukon Location, Yukon, Oklahoma
  - The Corvallis Clinic, Corvallis, Oregon
  - Summit Research, Portland, Oregon
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Velocity Clinical Research - Providence, Providence, Rhode Island
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - DelRicht Research, Charleston, South Carolina
  - Charleston Clinical Trials, LLC, Charleston, South Carolina
  - Velocity Clinical Research, Spartanburg, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Velocity Clinical Research- UNION, Union, South Carolina
  - Black Hills Center for American Indian Health, Rapid City, South Dakota
  - M3 Wake Research/ClinSearch, LLC, Chattanooga, Tennessee
  - Helios Clinical Research, Jackson, Tennessee
  - MultiSpeciality Clinical Research, Johnson City, Tennessee
  - Avant Reseach Associates, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - Tekton Research, LLC, Beaumont, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - 3A Research, LLC, El Paso, Texas
  - Helios, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - Helios Clinical Research, Houston, Texas
  - DM Clinical Research - CyFair, Houston, Texas
  - DM Clinical Research- Bellaire, Houston, Texas
  - Helios CR, Inc. Keller Tx, Keller, Texas
  - Research Your Health, Plano, Texas
  - DELRICHT RESEARCH at ZOMNIR FAMILY MEDICINE, Prosper, Texas
  - DM Clinical Research, San Antonio, Texas
  - IMA Clinical Research, San Antonio, Texas
  - Tekton Research Inc - San Antonio, San Antonio, Texas
  - San Marcos Family Medicine, San Marcos, Texas
  - Stephenville Medical & Surgical Clinic, PA, Stephenville, Texas
  - Breco Research - A Tarheel Clinical Research Site, Sugar Land, Texas
  - DM Clinical Research - Sugarland, Sugar Land, Texas
  - DM Clinical Research - Tomball, Tomball, Texas
  - DM Clinical Research, Tomball, Texas
  - Synexus Clinical Research US, Inc., Salt Lake City, Utah
  - CenExel - JBR, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - J. Lewis Research, Inc/Jordan River Family Medicine, South Jordan, Utah
  - Javara, Alexandria, Virginia
  - Velocity Clinical Research-Hampton, Hampton, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Velocity Clinical Research-Portsmouth, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Amherst Family Practice, Winchester, Virginia
  - Velocity Clinical Research- Spokane, Spokane, Washington
  - Confluence Health, Wenatchee, Washington
- Belgium (4):
  - Anima Research Center, Alken
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Sint Maarten, Mechelen
  - University of Antwerpen - Vaccinopolis, Wilrijk
- Bulgaria (16):
  - Medical center "Dr. Staykov" Ltd., Burgas
  - MHAT "Sveti Ivan Rilski", Kozloduy
  - Medical Center Medconsult Pleven, Lovech branch, Lovech
  - Medical Center Hera - Montana branch, Montana
  - MHAT "Dr. Stamen Iliev", Montana
  - Medical Center Medconsult Pleven, Pleven
  - AIPPMP Dr. Levena Kireva, Plovdiv
  - MHAT "Sv. Panteleymon" Ltd., Plovdiv
  - DCC-1 Sliven Lts., Sliven
  - MHAT Sliven to MMA Sofia, Sliven
  - Diagnostic & Consultancy Center Ascendent, Sofia, Sofia
  - Medical Center "Hera" EOOD, Sofia
  - Medical Center Excelsior - Base 2, Sofia
  - Medical Center Excelsior OOD, Base1, Sofia
  - Medical Centre "Sirtuin" Ltd, Sofia
  - AIPPMP D-r Zhaneta Demireva Ltd., Stamboliyski
- Canada (15):
  - Aviva Medical Diagnostics and Specialists Clinic and Heart & Vascular Centre, Burlington
  - CARe Clinic, Calgary, AB, Calgary
  - Centricity Research Quebec City, Lévis
  - Milestone Research Inc., London
  - Red Maple Trials, Ottawa
  - Centricity Research Pointe-Claire, Pointe-Claire
  - Clinique de Lebourgneuf, Québec
  - CARe , Red Deer, AB., Red Deer
  - Bluewater Clinical Research Group Inc., Sarnia
  - Stouffville Medical Research Institute, Stouffville
  - Canadian Phase Onward Inc., Toronto
  - Centricity Research Toronto LMC, Toronto
  - Diex Recherche, Trois-Rivières
  - Colchester Research Group, Truro
  - Diex Recherche Victoriaville, Victoriaville
- Estonia (5):
  - Vee Family Doctors' Center, Paide
  - Center of Clinical and Basic Research, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Innomedica OU, Tallinn
  - Clinical Research Center, Tartu
- Finland (5):
  - FVR - Finnish Vaccine Research Ltd - Espoo, Espoo
  - FVR - Finnish Vaccine Research Ltd - Kokkola, Kokkola
  - FVR - Finnish Vaccine Research Ltd - Oulu, Oulu
  - FVR - Finnish Vaccine Research Ltd - Tampere, Tampere
  - FVR - Finnish Vaccine Research Ltd - Järvenpää, Turku
- Georgia (6):
  - Unimed Adjara Ltd - Batumi Referral Hospital, Batumi
  - LTD "Hospital service", Kutaisi
  - LTD Clinic Rustavi, Rustavi
  - Emergency Cardiology Center named by acad. G. Chapidze, Tbilisi
  - Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - LTD Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
- Germany (21):
  - Emovis GmbH, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Velocity Clinical Research Berlin, GmbH, Berlin
  - Praxis Rinke, Bochum
  - Klinische Forschung Dresden GmbH, Dresden
  - Medizentrum Essen Borbeck, Essen
  - IKF Pneumologie, Frankfurt
  - Infektio Research GmbH & Co.KG, Frankfurt
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Velocity Clincial Research Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover Mitte GmbH, Hanover
  - Klinische Forschung Karlsruhe, Karlsruhe
  - SMO.MD, Magdeburg
  - Dermatologie Quist BAG Dres. Med. Quist Part G, Mainz
  - CDG Studienambulanz, München
  - Future meds Offenbach, Offenbach
  - Red-Institut, Oldenburg
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Studienzentrum Brinkum, Stuhr
  - Hautarztpraxis Leitz & Kollegen, Stuttgart
  - Velocity Clinical Research Wiesbaden, Wiesbaden
- South Korea (9):
  - Korea University Ansan Hospital, Ansan-si
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chungnam National University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsuing City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (28):
  - Panthera Biopartners site - York, Acomb, York
  - FutureMeds Birmingham, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Layton Medical Centre, Blackpool
  - Lakeside Healthcare, Corby
  - NHS Lothian - Western General Hospital, Edinburgh
  - Panthera Biopartners site - Enfield, Enfield
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - FutureMeds - Glasgow, Glasgow
  - Glasgow Panthera Biopartners Site, Glasgow
  - Barts Health NHS Trust - Mile End Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Guy's and St Thomas's NHS Foundation Trust, London
  - HMC Research Group, London
  - St George's University Hospitals (NHS Foundation Trust), London
  - Velocity Clinical Research - North London, London
  - Manchester University NHS Foundation Trust, Manchester
  - FutureMeds Wirral, Metropolitan Borough of Wirral
  - Infectious Diseases Research - Clinical Research Facility, Newcastle upon Tyne
  - Norfolk nand Norwich University Hospital, Norwich
  - University of Nottingham Health Service, Nottingham
  - Wansford Research Limited, Peterborough
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Portsmouth Hospitals University NHS Trust - Portsmouth Research Hub, Portsmouth
  - Panthera Biopartners - Manchester, Rochdale
  - Sheffield Panthera Biopartners Site, Sheffield
  - Southampton General Hospital, Southampton
  - Future Meds - Teesside, Stockton-on-Tees